CLINICAL TRIAL: NCT06196567
Title: The Effectiveness of Pulsed Electromagnetic Field Therapy on Muscle Strength and Function in Patients With End-stage of Knee Osteoarthritis Patients: a Randomized Controlled Trial
Brief Title: Pulsed Electromagnetic Field Therapy on Muscle Strength and Function in Patients With End-stage of Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Tim-Yun Michael ONG, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.210
Record Dates: First submitted 2023-12-08; First posted 2024-01-09 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; PEMF; Knee muscle strength; total knee replacement; knee pain and function
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three intervention groups, which will have treatment for 8 weeks prior to the surgery.
Who Masked: Investigator
Masking Description: It is single-blinded, the investigators don't know the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- active control group (Active Comparator): will receive the standard prehabilitation a physio-based exercise program designed to increase quadriceps muscle strength for 2 sessions per week for 8 weeks. Sessions will be performed at the same time (i.e., in the morning). The main programme comprised 5 sets of 10 repetitions for each exercise, with 60 rest between sets.
  Interventions: Other: exercise
- Pulsed Electromagnetic Field (PEMF) (Experimental): will receive the active PEMF treatment provided by a PEMF device (Quantum Tx, Singapore). Alternating leg will be exposed to PEMF for 10 minutes per session for 2 sessions per week for 8 weeks.
  Interventions: Device: PEMF
- standard prehabilitation plus PEMF intervention (Experimental): This group will have both the standard prehabilitation and PEMF intervention for 2 sessions a week for eight weeks.
  Interventions: Device: PEMF; Other: exercise

INTERVENTIONS:
Device: PEMF — Subjects will receive PEMF treatment with the duration of 8 weeks, twice a week with total 16 treatment sessions
  Arms: Pulsed Electromagnetic Field (PEMF); standard prehabilitation plus PEMF intervention
Other: exercise — do the exercise aimed at improving knee muscle strength,twice a week for 8 weeks before surgery
  Arms: active control group; standard prehabilitation plus PEMF intervention

SUMMARY:
End-stage OA knee is one of the most common musculoskeletal complaints, with over 34,000 patients waiting for joint replacement in Hong Kong and is expected to increase as the population continues to age constantly. The nominal waiting time for joint replacement in Hong Kong is long compared with many developed countries, averaging at 122 months, resulting in many elderly patients living with severe pain, limiting their daily activities. We are, therefore, in dire need to improve the well-being of this large and increasing group of patients as the capacity for operations remains limited.

It is important to maintain preoperative knee-extensor strength in the end-stage of knee OA awaiting TKR because the improvement of knee-extensor strength may postpone the need for surgery and increase the ability to perform functional activities after TKR at the same time.

PEMF exposure, on top of regular exercise training, may promote the secretion of myokine and in turn, promote muscle regeneration. These findings laid grounds for implementing PEMF treatment for end-stage knee OA patients to enhance muscle regeneration in periods with limited physical activity.

The novelty of this study is that this is the first RCT to examine if pulsed electromagnetic field therapy (PEMF), in addition to a standard rehabilitation, produces better muscle strength and functional performance before and after TKR in people with knee OA than either intervention alone. The impact of this study is particularly strong given end-stage patients waiting for knee replacement surgeries in Hong Kong.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is one of the most common chronic degenerative joint conditions affecting our ageing population. It is widely stated that OA is the leading cause of disability in elders due to discordant symptoms, such as pain and stiffness. Radiographic evidence of OA increased with age, from 8% in subjects younger than age 50, to over 60% in subjects aged 60 or above. Typically, conservative therapies that target symptoms are recommended as first- and second-line treatments for knee OA to reduce pain, stiffness, and activity limitations. However, when conservative therapies fail, they would then require total knee replacement (TKR). In 2022 to 2023, there were over 34,000 patients on the Hospital Authority (HA) waiting list for TKR. With only 3389 TKRs being performed, the nominal waiting time for TKR was outrageously long, 122 months in Hong Kong, as compared to an average of 9 months in Canada. Despite the efforts from the government to establish more joint replacement centres, the number of patients suffering from end-stage OA knees and requiring surgery will increase significantly as the population ages. Toward those requiring TKR, the excruciating pain would further cause significant functional impairment and lower health-related quality of life, which could eventually affect post-surgery outcomes. Although TKR appears to be an effective treatment in most people with end-stage Knee OA, 20%-40% of individuals remain dissatisfied. This is due to reduced leg strength occurring years after surgery, impaired functional capacity like poorer walking performance, greater deficits in physically demanding tasks such as stair climbing and poor performance of domestic duties .

The role of knee-extensor strength in the end-stage of Knee OA Knee-extensor muscle weakness has been regarded as a risk factor for knee OA. As shown, end-stage knee OA patients awaiting TKR had 35% reduced knee-extensor strength compared to healthy, age-matched individuals. In addition, pre-operative knee-extensor strength has also been found to be a predictor of postoperative functional ability up to a year following surgery. On average, patients would lose an additional 80% of their pre-operative knee-extensor strength shortly after TKA. Collectively, these data highlight the importance of maintaining preoperative knee-extensor strength in the end-stage of knee OA awaiting TKR and suggest that the improvement of knee-extensor strength may postpone the need for surgery and increase the ability to perform functional activities after TKR at the same time.

The role and limitation of prehabilitation before TKR The concept of preparing the body for a stressful event, such as surgery, has been named "prehabilitation". Prehabilitation was reported to positively affect knee OA symptoms and support patients' self-management of their knee OA condition, potentially postponing the need for surgery. As supported by the latest systematic review, it is important to focus on knee extensor muscle strength when evaluating the effects of prehabilitation before surgery in patients eligible for TKR. The review found that prehabilitation exercise could help to moderately increase knee extensor muscle strength and physical function and reduce pain. Moreover, a 30-40% increase in knee-extensor strength has been suggested to improve knee pain and disability. In conclusion, current prehabilitation has limited effects on improving sufficient knee extensor muscle strength.

Potential role of PEMF PEMF treatment utilizes a pulsed electromagnetic field to stimulate mitochondrial activity in skeletal muscle. Our group (Prof. Alfredo Franco-Obregon) showed that brief 10-minute exposure of 1 mT amplitude of PEMF (Quantum Tx) on myoblast in vitro could activate myogenesis. This can lead to a boost in repair and muscle regeneration via the release of myokines. Additionally, it plays an important role in regulating the production and secretion of myokine. Therefore, it is hypothesized that PEMF exposure, on top of regular exercise training, may promote the secretion of myokine and in turn promote muscle regeneration. These findings laid grounds to implement PEMF treatment for end-stage knee OA patients to enhance muscle regeneration in periods where limited physical activity is occurred. Also, this may help to set up a treatment regime for the PEMF device to impose myogenic effects, including exposure time per session, the number of treatment sessions and the duration of treatment.

Aims

The proposed project aims to set up a single-blinded randomized control trial to examine if pulsed electromagnetic field therapy (PEMF) in addition to a standard prehabilitation produces better muscle strength and functional performance before and after TKR in people with knee OA than either intervention alone.

To investigate the effect of PEMF in addition to a standard prehabilitation for muscle strength in end-stage OA knee patients.

To investigate the effect of PEMF in addition to a standard prehabilitation for knee symptoms and functional performance of OA knees in end-stage OA knee patients.

To investigate the effect of PEMF in addition to a standard prehabilitation for improving pain, function, and quality of life of OA knees in end-stage OA knee patients after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients end-stage knee OA over 50 waiting for TKR
* Patient has been scheduled for TKR at Prince of Wales Hospital
* Able to comply with the assessments and has given oral and written consent

Exclusion Criteria:

* Patients with connective tissue disorders or myositis condition
* History of any Hip & Knee joint replacement
* Patients with acute immobility (i.e., post hip fracture or post-acute hospital admission)
* Previous cases of any substances abuse
* Patients already had TKR for one knee before
* Patients are unable to transport themselves for intervention
* Patients have any neuromuscular or neurodegenerative conditions
* Patients have the history of inflammatory arthritis

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes of knee muscle strength | Day 0, 4th week, 8th week after the commencement the intervention and 6th week, 3 months, and 12 months after the TKR surgery
  The peak torque in kgf will be recorded with in 2 trials in the 5 seconds isometric muscle strength test.

SECONDARY OUTCOMES:
Appendicular muscle mass | Day 0, 4th week, 8th week after the commencement the intervention and 6th week, 3 months, and 12 months after the TKR surgery
  The appendicular muscle mass will tested using dual x-ray absorptiometry (DXA)
myokine evaluation-Brain-derived neurotrophic factor (BDNF) | Day 0, 8th week after the commencement the intervention and 6th week, 3 months, and 12th month after the TKR surgery
  Quantitative analysis for BDNF and proteins related to muscle metabolism will be performed by Human Myokine Magnetic Bead Panel (Millipore) with Bioplex-200 bead-based suspension assay system (LKSIHS core facilities), or enzyme-linked immunosorbent assay (ELISA) and report with pg/ml.
myokine evaluation-Fibroblast growth factor-21 (FGF-21) | Day 0, 8th week after the commencement the intervention and 6th week, 3 months, and 12th month after the TKR surgery
  Quantitative analysis for FGF-21 and proteins related to muscle metabolism will be performed by Human Myokine Magnetic Bead Panel (Millipore) with Bioplex-200 bead-based suspension assay system (LKSIHS core facilities), or enzyme-linked immunosorbent assay (ELISA) and report with pg/ml.
myokine evaluation-Interleukin-6 (IL-6) | Day 0, 8th week after the commencement the intervention and 6th week, 3 months, and 12th month after the TKR surgery
  Quantitative analysis for IL-6 and proteins related to muscle metabolism will be performed by Human Myokine Magnetic Bead Panel (Millipore) with Bioplex-200 bead-based suspension assay system (LKSIHS core facilities), or enzyme-linked immunosorbent assay (ELISA) and report with pg/ml.
myokine evaluation-Interleukin-15 (IL-15) | Day 0, 8th week after the commencement the intervention and 6th week, 3 months, and 12th month after the TKR surgery
  Quantitative analysis for IL-15 and proteins related to muscle metabolism will be performed by Human Myokine Magnetic Bead Panel (Millipore) with Bioplex-200 bead-based suspension assay system (LKSIHS core facilities), or enzyme-linked immunosorbent assay (ELISA) and report with pg/ml.
myokine evaluation-Irisin | Day 0, 8th week after the commencement the intervention and 6th week, 3 months, and 12th month after the TKR surgery
  Quantitative analysis for Irisin and proteins related to muscle metabolism will be performed by Human Myokine Magnetic Bead Panel (Millipore) with Bioplex-200 bead-based suspension assay system (LKSIHS core facilities), or enzyme-linked immunosorbent assay (ELISA) and report with pg/ml.
myokine evaluation-Insulin-like growth factor 1 (IGF-1) | Day 0, 8th week after the commencement the intervention and 6th week, 3 months, and 12th month after the TKR surgery
  Quantitative analysis for IGF-1 and proteins related to muscle metabolism will be performed by Human Myokine Magnetic Bead Panel (Millipore) with Bioplex-200 bead-based suspension assay system (LKSIHS core facilities), or enzyme-linked immunosorbent assay (ELISA) and report with pg/ml.
myokine evaluation-Insulin-Follistatin | Day 0, 8th week after the commencement the intervention and 6th week, 3 months, and 12th month after the TKR surgery
  Quantitative analysis for Follistatin and proteins related to muscle metabolism will be performed by Human Myokine Magnetic Bead Panel (Millipore) with Bioplex-200 bead-based suspension assay system (LKSIHS core facilities), or enzyme-linked immunosorbent assay (ELISA) and report with pg/ml.
myokine evaluation-Insulin-C- terminal of troponin T1 (TNNT1) | Day 0, 8th week after the commencement the intervention and 6th week, 3 months, and 12th month after the TKR surgery
  Quantitative analysis for TNNT1 and proteins related to muscle metabolism will be performed by Human Myokine Magnetic Bead Panel (Millipore) with Bioplex-200 bead-based suspension assay system (LKSIHS core facilities), or enzyme-linked immunosorbent assay (ELISA) and report with pg/ml.
Stair Ascent-Descent Assessment | Day 0, 4th week, 8th week after the commencement the intervention and 6th week, 3 months, and 12 months after the TKR surgery
  This test consisted of a stair climb, followed by a stair descent. The participants will begin from a standing start, and to be instructed to climb one flight (9 steps) of standard stairs by using the railing for balance if necessary. At the top of the stairs, they would immediately reverse in direction to descend from the same staircase. The time will be recorded. Less time means better function ability.
Chair Stand Test | Day 0, 4th week, 8th week after the commencement the intervention and 6th week, 3 months, and 12 months after the TKR surgery
  The chair stand test is a reliable test for assessment for low limb strength in patients. Patients will be asked to sit on a solid chair with arms on shoulders and feet with shoulder width apart. Time of 5 repetition will recorded.Less time means better function ability.
Postural Stability Assessment | Day 0, 4th week, 8th week after the commencement the intervention and 6th week, 3 months, and 12 months after the TKR surgery
  A force platform (Tekscan, U.S.) will be utilized to evaluate static postural control using the COP measures in static and dynamic postural control conditions. Sway path length of center of pressure (COP), velocity and ellipse area of COP will be recorded. These static postural conditions include stand on double leg with open and close eyes for 30s. The patients will perform two successful trials of each condition.
Short-Form 36 (SF-36) | Day 0, 4th week, 8th week after the commencement the intervention and 6th week, 3 months, and 12 months after the TKR surgery
  The SF-36 health survey uses 36 questions to measure a patient's functional health and well-being from a patient's point of view. It is a reliable and validated measure that summarises the patients' physical and mental health.higher score indicate a better outcome in each subscape.
Knee injury and Osteoarthritis Outcome Score | Day 0, 4th week, 8th week after the commencement the intervention and 6th week, 3 months, and 12 months after the TKR surgery
  Self-reported pain and physical function will be measured using the Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire. This 42-item questionnaire is divided into five subscales, which address pain, other disease symp¬toms, function in activities of daily living, function in sport and recreation, and quality of life. higher score indicate a better outcome in each subscape.
International Physical Activity Questionnaire (IPAQ) | Day 0, 4th week, 8th week after the commencement the intervention and 6th week, 3 months, and 12 months after the TKR surgery
  The IPAQ is a questionnaire that assesses and monitors a patient's physical activity and inactivity level. This instrument sums up a patient's activity level per week.
Visual Analogue Scale | Day 0, 4th week, 8th week after the commencement the intervention and 6th week, 3 months, and 12 months after the TKR surgery
  Severity of pain will be assessed using a visual analogue scale (VAS) which is a 10cm rating scale ranging from 'no pain at all' (score 0) to 'unbearable pain' (score 10). Patients will be instructed to mark a place on the horizontal line of the scale reflecting their knee pain severity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tim-Yun Ong, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Michael.Ong@Cuhk.Edu.Hk, Hong Kong, NEW Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 12 months after publication
Access Criteria: Journal reviewers